CLINICAL TRIAL: NCT02981147
Title: PEACe: Ivy, Thyme and Cisti Extract (Phytus) Efficacy in Acute Cough
Acronym: PEACe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE/PK/PYTUS/SP/2017-01
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2017-03

CONDITIONS: Cough; Common Cold
Keywords: cough; thyme; Cisti; Ivy Leaves
MeSH Terms: conditions — Cough; Common Cold | interventions — Phytotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Phytus (Cisti, thyme and Ivy leaves) given to patients on day 1 and day 4. On 4th day, night and day cough score along with adverse event will be assessed. Sponsor will bear the treatment cost during the study time period.
  Interventions: Drug: Phytus (Cisti, Thyme and Ivy Leaves)

INTERVENTIONS:
Drug: Phytus (Cisti, Thyme and Ivy Leaves) — Phytus is a medicinal herb containing Ivy leaves, Cisti and Thyme.
  Other Names: herbal medicine

SUMMARY:
The purpose of this study is to investigate the efficacy of Phytus in Acute Cough

DETAILED DESCRIPTION:
Common colds are the most frequently encountered human diseases worldwide. Common cold is a conventional term used for mild upper respiratory illnesses, which comprises a heterogeneous group of self-limited diseases caused by numerous viruses. The frequency is age-specific with fewer episodes in adults than in younger children. Cough due to the common cold is probably the most common cause of acute cough. In a significant subset of patients with "post infectious" cough, the etiology is probably an inflammatory response triggered by a viral upper respiratory infection (ie, the common cold). The resultant sub-acute or chronic cough can be considered to be due to an upper airway cough syndrome, previously referred to as postnasal drip syndrome.

Thyme leaf (Thymus vulgaris) expels phlegm and relieves congestion . It is antiseptic and an immune stimulant. The primary chemical constituents of Thyme include essential oil (borneol, carvacrol, cymol, linalool, thymol), bitter principle, tannin, flavonoids (apigenin, luteolin), saponins, and triterpenic acids. Thyme warms and stimulates the lungs, expels mucus, and relieves congestion. It also helps deter bacterial, fungal, and viral infections. The thymol content of thyme works as an expectorant and cough suppressant and is frequently used in cough syrups.

ELIGIBILITY:
Inclusion Criteria:

* Cough attributed to URTI such as the common cold
* Moderate to severe day cough according to questionnaire (score at least 3 on all 3 questions relating to day cough) considering the day prior to enrollment.
* Moderate to severe night cough score according to questionnaire (score at least 3 of 2 of the three questions relating to the evaluation of nocturnal cough

Exclusion Criteria:

* Diagnosis of chronic cardiac condition, or cystic fibrosis or any anatomical respiratory tract anomalies,
* Received antihistamines or any cough medicine the day prior to study entry,Known sensitivity to any component of Phytus

Ages: 2 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in day cough score at end of study | 4 nights (onset of trial Night 1 to Night 4)
  A validated cough questionnaire measuring 3 aspects of daytime cough (frequency, severity, bothersomeness) on a 7 point Likert scale was used each evening to rate the passed day, as regards these aspects. The scale rates each parameter from 0 (not at all) to 6 (extremely)

SECONDARY OUTCOMES:
Change in night cough score at end of study | 4 nights (onset of trial Night 1 to Night 4)
  A validated cough questionnaire measuring 5 aspects of night cough (frequency, severity, bothersomeness, child sleep and parents' sleep) on a 7 point Likert scale was used each morning to rate the past night. The scale rates each parameter from 0 (not at all) to 6 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Masood Jawaid, MRCS,FCPS, Study Director — PharmEvo Pvt Ltd
Locations (1):
- KCHS Medical Center 1st Floor, Tipu Sultan Road., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No